CLINICAL TRIAL: NCT00452244
Title: Randomized Phase II Trail Comparing Gefitinib Plus Simvastatin and Gefitinib Alone in Patients With Previously Treated Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Gefitinib With or Without Simvastatin in Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Ji-youn Han, Head, Center for Lung Cancer, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-06-177
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Lung Cancer
Keywords: Gefitinib; Simvastatin; NSCLC; Advanced NSCLC
MeSH Terms: conditions — Lung Neoplasms | interventions — Simvastatin; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- study arm (Experimental): Iressa (gefitinib) + simvastatin
  Interventions: Drug: simvastatin; Drug: gefitinib only
- control arm (Active Comparator): Iressa (gefitinib) only
  Interventions: Drug: gefitinib only

INTERVENTIONS:
Drug: simvastatin — Simvastatin 40mg/QD po daily every 3 weeks
  Other Names: simvarstar; IRESSA
  Arms: study arm
Drug: gefitinib only — gefitinib 250mg/QD po daily every 3 weeks
  Other Names: IRESSA

SUMMARY:
The epidermal growth factor receptor (EGFR) is a key regulator of growth, differentiation, and survival of epithelial cancers. In a small subset of tumors, the presence of activating mutations within the ATP binding site confers increased susceptibility to gefitinib, a potent tyrosine kinase inhibitor of EGFR. Agents that can inhibit EGFR function through different mechanisms may enhance gefitinib activity in patients lacking these mutations. Mevalonate metabolites play significant roles in the function of the EGFR; therefore, mevalonate pathway inhibitors may potentiate EGFR-targeted therapies. Targeting HMG-CoA reductase, the rate-limiting enzyme of mevalonate pathway, using lovastatin induces a potent apoptosis in a variety of tumor types. In an in vitro study, combining gefitinib and lovastatin treatment showed synergistic cytotoxic activity through enhanced inhibition of AKT activation by EGF in NSCLC and head & neck cancer cell lines. Therefore, the investigators would like to compare the combination effect of gefitinib and simvastatin, the specific and protein inhibitor of HMG-CoA reductase, with gefitinib alone in previously treated patients with NSCLC.

DETAILED DESCRIPTION:
Randomization

1. Sex (female vs. male)
2. ECOG PS (0/1 vs. 2/3)
3. Number of prior regimen (one vs. two).

Gefitinib (250 mg per day) + Simvastatin (40 mg per day) PO or Gefitinib (250 mg per day) alone

until progression or unacceptable toxicity

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologic diagnosis of NSCLC
2. Stage IV or selected stage IIIB (with positive pleural effusion or multiple ipsilateral lung nodules) according to the American Joint Committee on Cancer (AJCC).
3. Previously treated with at least one platinum-based chemotherapy.
4. Before study entry, a minimum of 21 days must have elapsed since any prior chemotherapy.
5. Prior radiation therapy is allowed as long as the irradiated area is not the only source of measurable disease.
6. No other forms of cancer therapy, such as radiation, immunotherapy for at least 2 weeks before the enrollment in study.
7. Performance status of 0-3 on the ECOG criteria.
8. At least one unidimensional measurable lesion meeting Response Evaluation Criteria in Solid Tumors (RECIST. 2000).- Estimated life expectancy of at least 8 weeks.
9. Patient compliance that allow adequate follow-up.
10. Adequate hematologic (ANC count ≥ 1,000/uL, platelet count ≥ 150,000/mm3), hepatic (bilirubin level≤1.5 mg/dL, AST/ALT ≤ 80 IU/L), and renal (creatinine concentration ≤ 1.5 mg/dL) function.
11. Informed consent from patient or patient's relative.
12. Males or females at least 18 years of age.
13. If female: childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of an approved contraceptive method (intrauterine device [IUD], birth control pills, or barrier device) during and for 3 months after trial. If male, use of an approved contraceptive method during the study and 3 months afterwards. Females with childbearing potential must have a urine negative hCG test within 7 days prior to the study enrollment.
14. No concomitant prescriptions including cyclosporin A, valproic acid, phenobarbital, phenytoin, ketoconazole.
15. Patients with brain metastasis are allowed unless there were clinically significant neurological symptoms or signs

Exclusion Criteria:

1. Presence of small-cell lung cancer alone or with NSCLC- Unresolved chronic toxic effects from previous anticancer therapy
2. Known severe hypersensitivity to gefitinib or any of the tablet excipients
3. Inability to swallow tablets
4. Other coexisting malignant disease (apart from basal-cell carcinoma)
5. More than three previous chemotherapy regimens for NSCLC
6. Previous treatment with an experimental agent of which the main mechanism of action is inhibition of epidermal growth factor receptor or its associated tyrosine kinase
7. Concomitant use of phenytoin, carbamazepine, rifampicin, barbiturates, or St John's wort; severe or uncontrolled systemic disease; clinically active interstitial lung disease (except uncomplicated lymphangitic carcinomatosis) pregnancy; and breastfeeding.
8. MI within preceding 6 months or symptomatic heart disease, including unstable angina, congestive heart failure or uncontrolled arrhythmia
9. Serious concomitant infection including post obstructive pneumonia
10. Major surgery other than biopsy within the past two weeks.
11. Pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2006-05; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Overall Response rate | every 8 weeks
  from C1D1 until confirmed disease progression

SECONDARY OUTCOMES:
Overall survival | every 12 weeks
  the first day of treatment to death
Toxicity | every 4 weeks
  From C1D1 to 1 months after the last dose adminitration
Pharmacogenetic and biomarker profile analysis | every 8 weeks
  From screening visit until confirmed disease progression
Time to progression | every 8 weeks
  From randomization date to disease progresssion or death date

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Youn Han, M.D.,Ph.D., Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Han JY, Kim JY, Lee SH, Yoo NJ, Choi BG. Association between plasma hepatocyte growth factor and gefitinib resistance in patients with advanced non-small cell lung cancer. Lung Cancer. 2011 Nov;74(2):293-9. doi: 10.1016/j.lungcan.2011.02.021. Epub 2011 Mar 26. PMID 21440951
- [Derived] Han JY, Lee SH, Yoo NJ, Hyung LS, Moon YJ, Yun T, Kim HT, Lee JS. A randomized phase II study of gefitinib plus simvastatin versus gefitinib alone in previously treated patients with advanced non-small cell lung cancer. Clin Cancer Res. 2011 Mar 15;17(6):1553-60. doi: 10.1158/1078-0432.CCR-10-2525. PMID 21411446